CLINICAL TRIAL: NCT02854111
Title: Using of Ice Cream for Diagnosis of Diabetes Mellitus and Impaired Glucose Tolerance
Brief Title: Using of Ice Cream for Diagnosis of Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Chutintorn Sriphrapradang, Assistant Professor, Ramathibodi Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-55-03
Record Dates: First submitted 2016-07-28; First posted 2016-08-03 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Ice Cream; Glucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- oral glucose tolerance test (Active Comparator): 75-g glucose A blood sample will be collected when the participants arrive. This is a fasting blood glucose value. Then the participants will be asked to drink a sweet liquid containing 75 g-glucose. Blood samples will be collected at timed intervals of 1 and 2 hours after you drink the glucose. This is a standard method for diagnosis of diabetes mellitus that called oral glucose tolerance test or OGTT.
  Interventions: Other: 75 g-glucose
- ice cream (Experimental): A blood sample will be collected when the participants arrive. This is a fasting blood glucose value. Then the participants will be asked to drink ice cream that contained carbohydrate 73.9 g. Blood samples will be collected at timed intervals of 1 and 2 hours after you eat the ice cream.
  Interventions: Other: ice cream

INTERVENTIONS:
Other: ice cream — The ice cream was made by nutritionists in Ramathibodi Hospital. It consisted of cornstarch, milk, sucrose, milk powder, egg yolk, and banana which contained carbohydrate 73.9 g, fat 27.7 g, protein 18.9 g for a total of 620.9 kcal with a cost of 35 bahts. The time for complete ingesting 75-g glucose and ice cream was 5 and 15 minutes, respectively.
  Arms: ice cream
Other: 75 g-glucose — The 75-g glucose is used for standard oral glucose tolerance test.
  Arms: oral glucose tolerance test

SUMMARY:
The overall global prevalence of type 2 diabetes mellitus (DM) is rising. Based on the latest Thai National Health Examination Survey, an estimated 3.2 million people had DM, of whom one-third was undiagnosed. The inexpensive oral glucose tolerance test (OGTT) is a more sensitive and reliable test of DM than fasting plasma glucose (FPG) or HbA1c, and is recommended for diagnosing DM and impaired glucose tolerance (IGT). Although the OGTT provides useful diagnostic information, poor patient tolerance of glucose solutions is inevitable.

DETAILED DESCRIPTION:
Regarding the diagnosis of DM, oral glucose tolerance test (OGTT) identifies about 2% more individuals than does fasting plasma glucose (FPG). Hence OGTT is the method that has high sensitivity compared to other methods for diagnosis of IGT (impaired glucose tolerance) and diabetes. However, standard OGTT with 75-g glucose has poor patient tolerance and might cause reactive hypoglycemia. The alternatives for 75-g glucose would help for screening of DM with better tolerance. There were previous studies investigated substitutes for oral glucose solution with cookies and muffin. In the present study we hypothesized that an alternative food such as ice cream, a favorite dessert, can use for evaluation of the diagnosis of DM and IGT instead of standard 75-g glucose.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer
* agree to participate by written informed consent

Exclusion Criteria:

* previous history of diabetes mellitus
* pregnant woman
* hospitalised patients
* underlying disease of liver and kidney disease
* who take any medications that interfere with plasma glucose levels such as steroid

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2013-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The correct diagnosis of diabetes mellitus | 2 hours
  We calculate the percentage of wrong diagnosis of diabetes mellitus when using ice cream instead of 75-g glucose (gold standard test). We also calculate sensitivity and specificity of ice cream test for diagnosis of diabetes mellitus.

SECONDARY OUTCOMES:
The correct diagnosis of impaired glucose tolerance | 2 hours
  We calculate the percentage of wrong diagnosis of impaired glucose tolerance using ice cream instead of 75-g glucose (gold standard test). We also calculate sensitivity and specificity of ice cream test for diagnosis of impaired glucose tolerance.

CONTACTS AND LOCATIONS:
Overall Officials: Chutintorn Sriphrapradang, M.D., Principal Investigator — Ramathibodi Hospital
Locations (1):
- Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chanprasertpinyo W, Bhirommuang N, Surawattanawiset T, Tangsermwong T, Phanachet P, Sriphrapradang C. Using Ice Cream for Diagnosis of Diabetes Mellitus and Impaired Glucose Tolerance: An Alternative to the Oral Glucose Tolerance Test. Am J Med Sci. 2017 Dec;354(6):581-585. doi: 10.1016/j.amjms.2017.08.007. Epub 2017 Aug 18. PMID 29208255